CLINICAL TRIAL: NCT06315686
Title: A Single-center Prospective Cohort Study to Explore the Efficacy and Prognosis of Dynamic Monitoring of Cerebrospinal Fluid ctDNA
Brief Title: The Dynamic Monitoring of Cerebrospinal Fluid ctDNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-ENDO-202209
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: NSCLC
MeSH Terms: interventions — Pemetrexed; aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Eligible patients with advanced non-small cell lung cancer with leptomeningeal metastasis were treated with vormetinib combined with OMMAYA lateral ventricle chemotherapy (pemetrexed).
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — The efficacy of Furmonertinib combined with OMMAYA lateral ventricle chemotherapy (pemetrexed) was evaluated once a week during the treatment phase. After the brain lesions were evaluated as CR, the drug holiday study phase was added. During the study period, the patients were followed up once a week until the investigators deemed the subjects unfit to continue to participate in the study or the efficacy was evaluated as disease progression (PD).
  Other Names: Furmonertinib

SUMMARY:
Focusing on advanced EGFR mutation in NSCLC patients with leptomeningeal metastasis, vormetinib combined with OMMAYA lateral ventricle chemotherapy (pemetrexed) was used to dynamically monitor ctDNA in cerebrospinal fluid (CSF), analyze the ctDNA gene mutation profile of CSF in different patients, and explore the relationship between ctDNA and efficacy and prognosis.

DETAILED DESCRIPTION:
This is a single-center prospective cohort study. Patients with advanced EGFR-mutated NSCLC with leptomeningeal metastasis were treated with vormetinib combined with OMMAYA lateral ventricle chemotherapy (pemetrexed). Dynamic monitoring of cerebrospinal fluid ctDNA was performed to analyze the ctDNA gene mutation profile of cerebrospinal fluid in different patients, and to explore the relationship between ctDNA and efficacy and prognosis. At the same time, the study of drug vacation in the treatment of leptomeningeal metastasis is to explore the efficacy and safety of brain drug vacation, so as to reduce the patient's tolerance to drugs and the side effects of drugs. The endpoint was progression-free survival (PFS) of intracranial lesions.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC patient with EGFR mutation, associated with leptomeningeal metastasis
* Patients who meet the requirements of OMMAYA cystlateral ventricle chemotherapy
* Age > 18 years
* Complete serologic tumor markers (CEA, SCC) and imaging data (enhanced CT and/or MRI, PET-CT)
* Liver, kidney, and hematologic measures were normal (as measured by laboratory testing within 1 week before enrollment in the absence of ongoing supportive care), with a neutrophil count of more than 1.5×109/L, a platelet count of more than 100×109/L, and a hemoglobin level of more than 9.0g/dl ，Bilirubin normal or <1.5×ULN; AST(SGOT), ALT(SGPT) <2.5×ULN; Serum creatinine <1.5×ULN
* The patients were fully aware of the study, provided voluntary written informed consent, and were able to adhere to the protocol-defined visit and follow-up procedures

Exclusion Criteria:

* Patients who do not meet the requirements of lateral ventricular chemotherapy
* History of allergy to vormetinib and pemetrexed
* Severe complications occurred during the treatment
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Severe infection in active stage or with poor clinical control
* Mentally ill, substance abusers and pregnant or lactating women
* No informed consent was signed
* Eligibility as judged by the other investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival time（PFS） | Up to 2 years
  The time from the initiation of treatment to the observation of disease progression or death from any cause.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 2 years
  Occurrence and severity of AEs by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: fang S cun, M.D., Study Director — Nanjing Brain Hospital
Locations (1):
- Nanjing Brain Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No